CLINICAL TRIAL: NCT05660954
Title: Biomarker Phase II Study Of Cabozantinib In Advanced Radioactive-Iodine Refractory Differentiated Thyroid Cancer.
Brief Title: Cabozantinib In Advanced Radioactive-Iodine Refractory Differentiated Thyroid Cancer.
Acronym: CABOTHYROID
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Collaborators: Ipsen (Industry); MFAR (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GETNE-T2216
Record Dates: First submitted 2022-12-02; First posted 2022-12-21 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Differentiated Thyroid Cancer
Keywords: Cancer; Thyroid; Cabozantinib
MeSH Terms: conditions — Neoplasms; Thyroid Diseases | interventions — cabozantinib

STUDY DESIGN:
Intervention Model Description: Experimental arm Patients with advanced radioactive-iodine refractory DTC who progressed to previous TKIs (including but not limited to lenvatinib or sunitinib). Patients will have not received previously cabozantinib, selective small-molecule BRAF kinase inhibitors, immune checkpoint inhibitor therapy, or systemic chemotherapy regimens
  All patients will receive cabozantinib at a fixed dose of 60 mg once a day (QD). Patients will continue study treatment until PD (either clinical or radiological), or until unacceptable toxicity, the need for another systemic anticancer treatment, or other reasons for treatment discontinuation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib, 60 mg (Experimental): Patients with advanced radioactive-iodine refractory DTC who progressed to previous TKIs (including but not limited to lenvatinib or sunitinib). Patients will have not received previously cabozantinib, selective small-molecule BRAF kinase inhibitors, immune checkpoint inhibitor therapy, or systemic chemotherapy regimens.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — * All enrolled patients will receive cabozantinib at a fixed dose of 60 mg once a day (QD). Patients will continue study treatment until PD (either clinical or radiological), or until unacceptable toxicity, the need for another systemic anticancer treatment, or other reasons for treatment discontinuation.
  * Patients will take the tablet(s) once daily at bed time except for Week 1 Day 1: the first dose of study treatment will be administered in the clinic so that each patient can be observed for initial tolerability. Subsequent doses will be self-administered at home. The tablets should be swallowed whole and not crushed and administered fasting for at least 2 hours before through 1 hour after. If a patient misses a dose, the missed dose should not be taken if it is less than 12 hours before the next dose.

SUMMARY:
CABOTHYROID is a prospective, exploratory, biomarker-focused, phase II, single-arm, non-randomized, non-blinded, investigator-initiated study of cabozantinib in patients with previously treated advanced radioactive-iodine refractory

DETAILED DESCRIPTION:
The trial will enroll competitively up to 41 subjects; male and female, ≥ 18 years, with ECOG PS 0-1 patients with advanced radioactive-iodine refractory differentiated thyroid cancer (DTC) who progressed to previous Tyrosine kinase inhibitors (TKIs), including but not limited to lenvatinib or sunitinib. Patients will have not received previously cabozantinib, selective small-molecule BRAF kinase inhibitors, immune checkpoint inhibitor therapy, or systemic chemotherapy regimens.

The design includes a screening phase in which patient eligibility is addressed, a treatment phase, and a follow-up phase.

Study treatment will begin as soon as possible after signing the informed consent and inclusion will be completed.

All patients will receive cabozantinib at a fixed dose of 60 mg once a day (QD). Patients will continue study treatment until PD (either clinical or radiological), or until unacceptable toxicity, the need for another systemic anticancer treatment, or other reasons for treatment discontinuation.

All patients will undergo periodic tumor assessments by CT or MRI scan every 12 weeks ± 14 days (3 months), and blood monitoring of tumor markers (i.e. thyroglobulin if applicable) every 12 weeks ± 3 days (2 months) from the start of study treatment until progression or patient withdrawal. Further CT/MRI scans could be performed upon suspicion of disease progression according to standard clinical practice and physician criteria. Safety will be assessed at every visit through continuous monitoring of signs and symptoms and periodic laboratory analysis.

The study includes the collection of two blood samples (baseline and after PD; 40 mL at each timepoint) for the determination of cf CHIP-seq (Chromatin immunoprecipitation-sequencing) and patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 18 years old.
2. Written informed consent approved by the Independent Ethics Committee (IEC), prior to the performance of any trial activities.
3. Histologically or cytologically confirmed diagnosis of DTC, including the following subtypes:

   (Note: results of a previous biopsy will be accepted):
   1. Papillary thyroid carcinoma (PTC) including histological variants of PTC such as follicular variant, tall cell, columnar cell, cribriform-morular, solid, oxyphil, Warthin-like, trabecular, tumor with nodular fasciitis-like stroma, Hürthle cell variant of papillary carcinoma, poorly differentiated.
   2. Follicular thyroid carcinoma (FTC) including histological variants of FTC such as Hürthle cell, clear cell, insular, and poorly differentiated.
4. Measurable disease according to RECIST 1.1 on computed tomography/magnetic resonance imaging (CT/MRI) performed within 28 days prior to first dose of study treatment.
5. Must have been previously treated with or deemed ineligible for treatment with Iodine-131 for DTC.
6. Must have been previously treated and experienced documented radiographic progression per RECIST 1.1 with one or two of the following vascular endothelial growth factor (VEGF) targeting TKI agents for DTC:

   1. Lenvatinib first-line or,
   2. Sorafenib first-line or,
   3. Two prior vascular endothelial growth factor receptor (VEGFR) TKIs.
7. Recovery to baseline or ≤ Grade 1 (Common Terminology Criteria for Adverse Events Version 5 [CTCAE v 5.0]) from toxicities related to any prior treatments, unless AEs are clinically nonsignificant and/or stable on supportive therapy.
8. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.
9. Adequate organ and bone marrow function based upon meeting all of the following laboratory criteria within 10 days before first dose of study treatment:

   1. Absolute neutrophil count ≥ 1500/mm3 (≥ 1.5 GI/L) without receipt of granulocyte colony-stimulating factor support within 2 weeks before screening laboratory sample collection.
   2. Platelets ≥ 100,000/mm3 (≥ 100 GI/L) without receipt of transfusion within 2 weeks before screening laboratory sample collection
   3. Hemoglobin ≥ 9 g/dL (≥ 90 g/L) without receipt of transfusion within 2 weeks before screening laboratory sample collection
   4. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 3 × upper limit of normal (ULN). ALP ≤ 5 × ULN if the subject has documented bone metastases
   5. Bilirubin ≤ 1.5 × the upper limit of normal (ULN). For subjects with known Gilbert's disease ≤ 3 × ULN
   6. Serum creatinine ≤ 2.0 × ULN or calculated creatinine clearance ≥ 30 mL/min (≥ 0.5 mL/sec) using the Cockcroft-Gault
   7. Urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol)
10. Female subjects of childbearing potential (WOCBP) must provide a negative urine pregnancy test at screening, and must agree to use a medically accepted and highly effective birth control method (i.e. those with a failure rate less than 1%; for the duration of the study treatment and for 4 months after the final dose of cabozantinib.

    - A woman is considered of childbearing potential ( i.e. fertile) following menarche and until becoming post-menopausal unless permanently sterile. Women will be considered post-menopausal if they have been amenorrhoeic for 12 months without an alternative medical cause. The following age-specific requirements apply:
    1. Amenorrheic for ≥1 year in the absence of chemotherapy and/or hormonal treatments
    2. Luteinizing hormone (LH) and/or follicle stimulating hormone and/or estradiol levels in the post-menopausal range
    3. Radiation induced oophorectomy with last menses >1 year ago
    4. Chemotherapy induced menopause with >1 year interval since last menses
    5. Surgical sterilization (bilateral oophorectomy or hysterectomy)
    6. Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
    7. Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
11. Non-sterile males must be willing to use a highly effective method of birth control for the duration of the study treatment and for 4 months after the final dose of cabozantinib.

    A sterile male is defined as:
    1. One for whom azoospermia has been previously demonstrated in a semen sample examination as definitive evidence of infertility.
    2. Males with known "low sperm counts" (consistent with "sub-fertility") are not to be considered sterile for purposes of this study.
12. Capable of understanding and complying with the protocol requirements and signed informed consent.

Exclusion Criteria:

1. Prior treatment with any of the following:

   1. Cabozantinib.
   2. Selective small-molecule BRAF kinase inhibitor (eg, vemurafenib, dabrafenib).
   3. Immune checkpoint inhibitor therapy (eg, PD-1 or PD-L1 targeting agent).
   4. Systemic chemotherapy regimen (given as a single agent or in combination with another chemotherapy agent).
2. Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks or 5 half-lives of the agent, whichever is longer, before first dose of study treatment.
3. Receipt of any type of anticancer antibody (including investigational antibody) within 4 weeks before first dose of study treatment.
4. Receipt of radiation therapy for bone metastasis within 2 weeks or any other radiation therapy within 4 weeks before first dose of study treatment. Patients with clinically relevant ongoing complications from prior radiation therapy that have not completely resolved are not eligible (eg, radiation esophagitis or other inflammation of the viscera).
5. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of inclusion.
6. Concomitant anticoagulation with oral anticoagulants (eg, warfarin, direct thrombin and Factor Xa inhibitors) or platelet inhibitors (eg, clopidogrel), except for the following allowed anticoagulants:

   1. Low-dose aspirin for cardioprotection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
   2. Anticoagulation with therapeutic doses of LMWH in subjects without known brain metastases who are on a stable dose of LMWH for at least 6 weeks before first dose of study treatment and who have had no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
7. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

   a. Cardiovascular disorders: i. Congestive heart failure class 3 or 4 as defined by the New York Heart Association, unstable angina pectoris, serious cardiac arrhythmias.

   ii. Uncontrolled hypertension defined as sustained BP > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment.

   iii. Stroke (including transient ischemic attack [TIA]), myocardial infarction, or other ischemic event, or thromboembolic event (eg, deep venous thrombosis [DVT], pulmonary embolism) within 6 months before first dose of study treatment. Note: Patients with a more recent diagnosis of DVT are allowed if stable, asymptomatic, and treated with LMWH for at least 6 weeks before first dose of study treatment.

   b. Gastrointestinal disorders (eg, malabsorption syndrome or gastric outlet obstruction) including those associated with a high risk of perforation or fistula formulation: i. Tumors invading the GI tract, active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic or biliary duct, or gastric outlet obstruction.

   ii. Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose of study treatment. Note: Complete healing of an intra-abdominal abscess must be confirmed prior to the first dose of study treatment.

   c. Clinically significant hematemesis or hemoptysis of > 0.5 teaspoon (> 2.5 mL) of red blood or history of other significant bleeding within 3 months before the first dose of study treatment.

   d. Cavitating pulmonary lesion(s) or known endobronchial disease manifestation. e. Lesions invading major pulmonary blood vessels. f. Other clinically significant disorders such as: i. Active infection requiring systemic treatment, infection with human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome-related illness, or chronic hepatitis B (HBV) or C (HCV) infection.

   ii. Serious non-healing wound/ulcer/bone fracture. iii. Malabsorption syndrome. iv. Moderate to severe hepatic impairment (Child-Pugh B or C). v. Requirement for hemodialysis or peritoneal dialysis. vi. Uncontrolled diabetes mellitus. vii. History of solid organ transplantation.
8. Major surgery (eg, GI surgery, removal or biopsy of brain metastasis) within 8 weeks before the first dose of study treatment. Complete wound healing from major surgery must have occurred 4 weeks before the first dose of study treatment and from minor surgery (eg, simple excision, tooth extraction) at least 10 days before the first dose of study treatment. Patients with clinically relevant ongoing complications from prior surgery are not eligible.
9. Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 28 days before the first dose of study treatment.

   Note: If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these 3 consecutive results for QTcF will be used to determine eligibility.
10. Patients who are not able to swallow tablets.
11. Previously identified allergy or hypersensitivity to components of the study treatment formulations.
12. Diagnosis of another malignancy within 3 years before the first dose of study treatment, except for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy.
13. Women pregnant or breastfeeding. Fertile and sexually active patients who are not willing to use the appropriate highly effective contraceptive methods.
14. Any underlying medical or psychiatric disorder, which, in the opinion of the investigator, makes the administration of cabozantinib unsafe or interferes with the informed consent process or trial procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Gene expression of molecular biomarkers characteristics of the pathology | Time point: At baseline, before any dose of study treatment
  Gene expression levels in the sample will be reported as media and interquartile range for each one of the biomarkers included in the determination. Determination of the expression of the molecular markers will perform applied chromatin immunoprecipitation of cell-free nucleosomes carrying active chromatin modifications followed by sequencing chromatin immunoprecipitation (cfChIP-seq) in blood samples. A blood sample of each patient will be collected for cfChIP-seq analysis in the baseline, before any dose of study treatment (week0)
Gene expression of molecular biomarkers characteristics of the pathology | Time point: Throughout the study period, approximately 2 years per patient
  Gene expression levels in the sample will be reported as media and interquartile range for each one of the biomarkers included in the determination. Determination of the expression of the molecular markers will perform applied chromatin immunoprecipitation of cell-free nucleosomes carrying active chromatin modifications followed by sequencing chromatin immunoprecipitation (cfChIP-seq) in blood samples. A blood sample of each patient will be collected and cfChIP-seq test will be performed as soon as the patient progresses according to RECIST 1.1 guidelines

SECONDARY OUTCOMES:
Objective response rate (ORR) | Throughout the study period, approximately 2 years per patient
  Objective response rate (ORR), primary endpoint for efficacy: Assessed by the investigator through imaging follow-up (CT scan/MRI) using RECIST 1.1. This will be considered as the percentage/proportion of patients with confirmed complete response (CR) or partial response (PR) as their overall best response throughout the study period. Objective responses will be assessed locally by the investigator according to RECIST, version 1.1, and indicating the change in size of tumors as compared with baseline, at the first dose of study treatment.
Disease control rate (DCR) | Throughout the study period, approximately 2 years per patient
  Percentage/proportion of patients with complete response (CR) or partial response (PR), according to ORR definition for the trial, or maintained stable disease (SD) as their overall best response, assessed by imaging follow-up (CT scan/MRI) and RECIST 1.1 criteria. Stable disease should be maintained for at least 4 months to be considered as a Chemical, Biological, or Radiological (CBR) event
Duration of response (DoR) | Throughout the study period, approximately 2 years per patient
  DoR is defined as the time from first confirmed response (CR or PR), according to ORR definition for the trial, to the date of the documented PD as determined using RECIST 1.1 criteria or death due to any cause, whichever occurs first. Those patients with response and without PD or death event will be censored on the date of their last tumor assessment.
Progression-free survival (PFS) | Throughout the study period, approximately 2 years per patient
  PFS is defined as time from first dosing date to the date of confirmed PD according to RECIST 1.1. Patients alive and free of events at the date of the analysis will be censored at their last known tumor assessment. Patients who start a new treatment line without progression will be censored on the date of first dose of the subsequent anticancer treatment.
Overall survival (OS) | Throughout the study period, approximately 2 years per patient
  Defined as the time elapsed from the first dose of study treatment until death from any cause. We will assess the median OS, estimated by Kaplan-Meier. Patients alive and free of events at the date of the analysis will be censored at their last known contact. Survival will be assessed by recording patient status at each visit according to Table 1. Long term follow up to be performed at least every 6 months.
Frequency of Adverse events (AEs) leading to treatment discontinuation. | Throughout the study period, approximately 2 years per patient
  Percentage of patients experiencing an adverse event leading to discontinuation of treatment
Health-related quality of life (HRQoL), assessed through the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30) version 3. | Throughout the study period, approximately 2 years per patient
  The EORTC QLQ-C30 questionnaire is a specific questionnaire validated for cancer that is composed of 30 questions or items. The questionnaire is structured in 5 functional scales (physical functioning, daily activities, emotional functioning, cognitive functioning and social functioning), 3 symptom scales (fatigue, pain and nausea, vomiting), 1 global health status scale, and 6 independent items (dyspnea, insomnia, anorexia, constipation, diarrhea and economic impact). Values between 1 and 4 (1: not at all, 2: a little, 3: quite, 4: a lot) are assigned according to the patient's responses to the item, only in items 29 and 30 are they evaluated with a score of 1 to 7 (1: dreadful, 7: excellent). The scores obtained are standardized and a score between 0 and 100 is obtained, which determines the level of impact of the cancer on the patient on each of the scales. A higher score indicating a better HRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Jaume Capdevila, M.D; PhD, Study Chair — Hospital Vall d'Hebron
Locations (9):
- Spain (9):
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Complejo Asistencial Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) anonymized could be shared upon request if the use is within the scope and protection level authorized by the patients by the signature of the informed consent